CLINICAL TRIAL: NCT05816889
Title: Investigation of Exercise Capacity, Muscle Oxygenation and Physical Activity Level in Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 35
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Upper extremity exercise capacity (6 minutes pegboard and ring test), muscle oxygenation ("moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), physical activity level (multi-sensor activity monitor) and fatigue (Parkinson's fatigue scale) will be evaluated.
- Healthy Controls: Upper extremity exercise capacity (6 minutes pegboard and ring test), muscle oxygenation ("moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), physical activity level (multi-sensor activity monitor) and fatigue (Parkinson's fatigue scale) will be evaluated.

SUMMARY:
The primary aim of this study is to compare maximum and functional exercise capacity and muscle oxygenation during exercise test in patients with Parkinson's disease. The secondary aim is to evaluate respiratory functions, respiratory muscle strength and endurance, peripheral muscle strength, physical activity level, shortness of breath and fatigue in Parkinson's patients and compare with healthy individuals.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common neurodegenerative disease. The main motor symptoms in Parkinson's disease are tremor, rigidity, bradykinesia, and decreased postural reflexes, and respiratory problems are seen that cause mortality. Disturbances in the control of the epiglottis, laryngeal and pharyngeal muscles may cause aspiration pneumonia. The coughing or exhalation reflex requires coordinated motor activity and inadequate airway defense poses a risk for pneumonia. Upper airway obstruction may occur due to rigidity and fatigue in the thyroarytenoid muscles. It can cause a decrease in lung volumes and thus the development of restrictive respiratory function abnormality.

Pulmonary functions, exercise capacity, respiratory muscle strength and endurance, peripheral muscle strength, physical activity level and fatigue were affected in patients. The number of studies on these subjects is limited.

Mitochondrial dysfunction in Parkinson's patients has been proven in several studies. There is no study in the literature evaluating muscle oxygenation at rest and during exercise in Parkinson's patients.

The primary aim of this study is to compare maximum and functional exercise capacity and muscle oxygenation during exercise test in patients with Parkinson's disease. The secondary aim is to evaluate respiratory functions, respiratory muscle strength and endurance, peripheral muscle strength, physical activity level, shortness of breath and fatigue in Parkinson's patients and compare with healthy individuals.

The study was planned cross-sectional. Patients with Parkinson Disease referred to the Cardiopulmonary Rehabilitation Unit of Gazi University Physiotherapy and Rehabilitation Department by the physicians of the Neurology Department of Gazi University Faculty of Medicine will be included in the study. At least 26 patients with Parkinson Disease and at least 26 healthy controls of similar age and sex will be evaluated in the study. The assessments will be completed in two days.

Upper extremity exercise capacity (6 minutes Pegboard and Ring Test), muscle oxygenation ("Moxy" monitor), functional exercise capacity(6 minutes walk test), respiratory functions (spirometer), respiratory muscle strength (mouth pressure measurement), respiratory muscle endurance (incremental threshold loading test), peripheral muscle strength (dynamometer), physical activity level (multi-sensor activity monitor) and fatigue (Parkinson's Fatigue Scale) will be evaluated.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria for Patients:

1. Between the ages of 45-80
2. Diagnosed with Parkinson's disease
3. Volunteer to participate in the study

Inclusion Criteria for Healthy Controls:

1. Healthy adults aged 45-80 years
2. Volunteer to participate in the study

Exclusion Criteria:

Exclusion Criteria for Patients:

1. Having a neurological disease other than Parkinson's disease
2. Having a diagnosed lung disease that may affect respiratory functions
3. Having had Coronavirus disease (COVID-19)
4. Have a smoking history of at least 10 pack×years or more.
5. Those with absolute and relative contraindications to exercise tests according to the American College of Sports Medicine (ACSM)
6. Those with a Mini Mental State Rating Scale score less than 18
7. Having orthopedic, neurological or psychological problems that would limit evaluations

Exclusion Criteria for Healthy Controls:

1. Those with a Mini Mental State Rating Scale score less than 18
2. Have a smoking history of at least 10 pack years or more.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 26 patients with Parkinson's diseasewill be included in patients group and 26 healthy individuals will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Lower extremity exercise capacity | First Day
  Lower extremity exercise capacity will be evaluated with six- minute walking test. The test will be performed according to the criteria of the American Thoracic Society and the European Respiratory Society.
Upper extremity exercise capacity | Second Day
  Upper extremity exercise capacity will be evaluated with the six-minute pegboard and ring test (6-PBRT). A pegboard with two upper and lower bars set at participants shoulder level and above the shoulder level will used. Ten rings will placed on both the lower bars. Patients will be asked to move a single ring at a time with both hands from the lower bars to the upper. The score is the total number of rings moved the six-minute period.
Muscle Oxygenation | First and Second Day
  Muscle oxygenation assessment will be performed using the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device will be placed on the 1/3 lower motor point of the quadriceps muscle group of the dominant leg and on the dominant arm deltoid muscle. A minimum of 3 minutes will be waited until the resting measurements and skeletal muscle oxygenation (StO2) signal stabilize. The measurements will be repeated during six minute walking test and six minute pegboard and ring test.

SECONDARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be measured with a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria.
Respiratory muscle endurance | Second Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load. The test will be started with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80% and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period will be recorded.The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Pulmonary function (Forced vital capacity (FVC) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced vital capacity (FVC) will be measured.
Pulmonary function (Forced expiratory volume in the first second (FEV1) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. FEV1 / FVC will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Peak flow rate (PEF) will be measured.
Muscle Strength | First Day
  Peripheral muscle strength will be evaluated with a dynamometer.
Physical activity (Total energy expenditure) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Fatigue | Second Day
  Fatigue will be evaluated using the Parkinson Fatigue Scale. Total score varies between 16-80. As the score increases, the severity of fatigue increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur GÜVENİR, Pt., Study Chair — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Ece BAYTOK, MSc, Principal Investigator — Gazi University; Betül YOLERİ, MSc, Principal Investigator — Gazi University; Ayşe BORA TOKÇAER, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No